CLINICAL TRIAL: NCT06386523
Title: Standardization of a New Psychophysical Olfactory Test, TODA2
Acronym: TODA-STAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-AOI-03
Record Dates: First submitted 2024-04-19; First posted 2024-04-26 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Patients Without an Olfactory Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Passage of olfactory tests (Experimental): Passage of olfactory tests: TODA2 and Sniffin Stick Test
  Interventions: Diagnostic Test: Passage of olfactory tests

INTERVENTIONS:
Diagnostic Test: Passage of olfactory tests — test TODA2 and Sniffin Stick Test

SUMMARY:
Recruitment of patients consulting the IUFC for another pathology unrelated to an olfactory disorder:

Interview and clinical examination and Passing the 2 olfactory tests for 30 voluntary's patients, a second consultation of 15 minutes including the time of the test within 7 days after the 1st

DETAILED DESCRIPTION:
Recruitment of patients consulting the IUFC for another pathology unrelated to an olfactory disorder (otosclerosis, pre- surgery, tonsillectomy, cosmetic surgery)

Data collection methods: 2 parts (duration approximately 1.5 hours) and for 30 volunteer patients, a second consultation of 15 minutes including the time of the test within 7 days after the 1st:

1. Interview and clinical examination
2. Passage of olfactory tests: TODA2 and Sniffin Stick Test in unirhinal
3. On a voluntary basis, and within a limit of 30 patients, those who agree to come back a second time will be able to benefit from a second pass of the TODA2 on Day 7.

ELIGIBILITY:
Inclusion Criteria:

* Subjects > 18 years old
* No olfactory complaints; subjective estimation of "normal" olfaction
* Affiliated to the Social Security system
* Signing of informed consent

Exclusion Criteria:

* Parosmia/phantosmia, hyposmia/anosmia, pre-existing subjective dysgeusia/ageusia
* ATCD of sinus or cranial neoplasia
* ATCD of sinus or cranial radiotherapy
* Neurological or neurodegenerative disease
* ATCD of persistent post-viral hyposmia or anosmia (including COVID) (more than 3 months)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Passage of olfactory tests: | Day 0
  TODA2
Passage of olfactory tests: | Day 0
  Sniffin Stick Test
Passage of olfactory tests: | Day 7
  TODA2

SECONDARY OUTCOMES:
Identify confounding factors, i.e. factors that can influence the results of the olfactory test | Day 0
  gender of patients
Identify confounding factors, i.e. factors that can influence the results of the olfactory test | Day 0
  Age of patients

CONTACTS AND LOCATIONS:
Overall Officials: Clair VANDERSTEEN, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (2):
- France (2):
  - CH de Cannes, Cannes
  - CHU de Nice, Nice

IPD SHARING:
Plan to Share IPD: No